CLINICAL TRIAL: NCT04040413
Title: Institutional Bariatric Database Registry
Brief Title: Database Maintenance for Bariatric Procedures
Status: Recruiting | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, David Goitein MD, Head, Bariatric and Metabolic Surgery, Sheba Medical Center
Other Study IDs: SMC-14-1828
Record Dates: First submitted 2019-07-26; First posted 2019-07-31 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Obesity, Morbid; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bariatric surgery — All bariatric procedures

SUMMARY:
Bariatric surgery registry for quality control and investigational purposes.

ELIGIBILITY:
Inclusion Criteria:

* morbid obesity

Exclusion Criteria:

* unfit for surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All morbidly obese individuals seeking bariatric surgery and approved by multidisciplinary bariatric committee.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Surgery type | 10 years
  Sleeve gastrectomy or Roux-Y gastric bypass (RYGBP) or Single anastomosis gastric bypass (SAGB) or biliopancreatic diversion (BPD/DS) or single anastomosis duodeno-ilial bypass (SADI)
Percent total weight loss (%TWL) | 1 year from surgery
  [(Weight at time of surgery - Weight at time point)/Weight at time of surgery]X100
Percent total weight loss (%TWL) | 5 years from surgery
  [(Weight at time of surgery - Weight at time point)/Weight at time of surgery]X100
Percent total weight loss (%TWL) | 10 years from surgery
  [(Weight at time of surgery - Weight at time point)/Weight at time of surgery]X100
Percent BMI loss (%BMIL) | 1 year from surgery
  [BMI at time of surgery - BMI at time point)/BMI at time of surgery] X 100
Percent BMI loss (%BMIL) | 5 years from surgery
  [BMI at time of surgery - BMI at time point)/BMI at time of surgery] X 100
Percent BMI loss (%BMIL) | 10 years from surgery
  [BMI at time of surgery - BMI at time point)/BMI at time of surgery] X 100

SECONDARY OUTCOMES:
Co-morbidity resolution | 1 year from surgery
  Cessation of medication/s used to treat weight-related co-morbidities (i.e. diabetes mellitus type 2, hypertension, dyslipidemia, degenerative joint disease etc.)
Co-morbidity resolution | 5 years from surgery
  Cessation of medication/s used to treat weight-related co-morbidities (i.e. diabetes mellitus type 2, hypertension, dyslipidemia, degenerative joint disease etc.)
Co-morbidity resolution | 10 years from surgery
  Cessation of medication/s used to treat weight-related co-morbidities (i.e. diabetes mellitus type 2, hypertension, dyslipidemia, degenerative joint disease etc.)
30 day morbidity/mortality | up to 30 days from intervention
  30 day morbidity/mortality according to Clavien Dindo criteria
long-term morbidity/mortality | 31 days to 10 years from surgery
  morbidity/mortality according to Clavien Dindo criteria after 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No